CLINICAL TRIAL: NCT07008898
Title: Sequence of Midurethral Sling Placement During Robotic Sacrocolpopexy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Gabriela Halder, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 300014707
Record Dates: First submitted 2025-05-27; First posted 2025-06-06 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Stress Incontinence Female; Pelvic Organ Prolapse
Keywords: Stress incontinence; Pelvic organ prolapse; Midurethral sling; Sucess rates; Complication rates; Patient satisfaction
MeSH Terms: conditions — Pelvic Organ Prolapse; Urinary Incontinence, Stress; Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Midurethral sling placed before robotic sacrocolpopexy (Active Comparator): Midurethral sling placed after robotic sacrocolpopexy
  Interventions: Procedure: Midurethral sling placed before robotic sacrocolpopexy
- Midurethral sling placed after robotic sacrocolpopexy (Active Comparator)
  Interventions: Procedure: Midurethral sling placed after robotic sacrocolpopexy

INTERVENTIONS:
Procedure: Midurethral sling placed before robotic sacrocolpopexy — Sequence of midurethral sling placement (before or after suspension of the vaginal apex) during robotic sacrocolpopexy is largely surgeon-dependent and dictated by training and experience. This study will examine whether there are any differences in continence and patient satisfaction between patients in whom slings are placed prior to suspension of the vaginal apex during robotic sacrocolpopexy versus after.
  Arms: Midurethral sling placed before robotic sacrocolpopexy
Procedure: Midurethral sling placed after robotic sacrocolpopexy — Sequence of midurethral sling placement (before or after suspension of the vaginal apex) during robotic sacrocolpopexy is largely surgeon-dependent and dictated by training and experience. This study will examine whether there are any differences in continence and patient satisfaction between patients in whom slings are placed prior to suspension of the vaginal apex during robotic sacrocolpopexy versus after.
  Arms: Midurethral sling placed after robotic sacrocolpopexy

SUMMARY:
This study looks at the best time to place a midurethral sling (MUS), which is a small piece of mesh used to treat stress urinary incontinence (SUI) (leaking urine when you cough, laugh, or exercise). The sling is placed during a type of surgery called robotic sacrocolpopexy (RSC). This surgery helps fix pelvic organ prolapse, when organs like the bladder or uterus drop from their normal place.

Doctors can place the sling either before or after they lift and support the top of the vagina during surgery, but they aren't sure which timing works better. In this study, investigators are comparing what is the best time to place the sling, how the patient feels after surgery and if a patient's symptoms got better or worse.

DETAILED DESCRIPTION:
Investigators will conduct a prospective, randomized, noninferiority trial on patients undergoing retropubic midurethral sling (RP MUS) placement at the time of robotic-assisted sacrocolpopexy (RSC).

Patients scheduled to undergo retropubic midurethral sling placement at the time of robotic- assisted sacrocolpopexy will be invited to participate during regularly scheduled preoperative visits with their urogynecologic provider. Participants will be randomized to receive RP MUS before RSC or after RSC. Randomization will be conducted in RedCap. Randomization will be performed using a variable permutated block randomization scheme. The Randomization window will be +/- 4 days before their scheduled surgery, and patients will be blinded to sequence of MUS placement intraoperatively.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Able to speak and read English and Spanish

  * Diagnosis of pelvic organ prolapse stage 2-4
  * Planning to undergo a robotic-assisted sacrocolpopexy
  * Demonstrable SUI (either by CST, with or without prolapse reduction, or UDS) within the year prior to enrollment
  * Planning to undergo concomitant SUI correction with MUS at the time of RSC

Exclusion Criteria:

* Less than 18 years of age
* Unable to speak and read English or Spanish
* No diagnosis of SUI (prophylactic slings)
* History of prior surgery for SUI
* Bladder capacity <200 mL or post-void residual (PVR) >150 mL
* Current genitourinary fistula or urethral diverticulum

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Urinary Distress Index, Short Form (UDI-6) scores at 3 months postoperative | 3 months
  The primary outcome will be change between baseline and 3 months stress urinary incontinence symptoms as measured by the UDI-6. Scores for the UDI-6 range from 0 to 100 has an MCID of 5.8, with higher scores indicating worse symptoms.

SECONDARY OUTCOMES:
Provocative stress test results at 6 weeks postoperative | 6 weeks
  Patients will be examined in the office during 6-week postoperative visit as is routine practice and assess for leakage of urine during empty supine provocative cough stress test.
Need for re-treatment for stress urinary incontinence (SUI) at 6 weeks postoperative | 6 weeks
  If recurrent stress urinary incontinence is noted to be present at 6-weeks postoperative, whether or not patients elect to proceed with additional treatment will be assessed.
Change in total Pelvic Organ Prolapse/Incontinence Sexual Questionnaire (PISQ-IR) at 3 months postoperative | 3 months
  PISQ-IR will be administered at enrollment and at 3 months postoperative, and scores will be compared.
Change in total Incontinence Impact Questionnaire, Short Form (IIQ-7) scores at 3 months postoperative | 3 months
  IIQ-7 will be administered to patients at enrollment and at 3 months postoperative, and scores at these two time points will be compared.
Complications (graded as Clavien Dindo) | 6 weeks
  Complications occurring during or after concomitant RSC and RP MUS will be recorded between both groups and compared.
Objective surgical data such as operative time | 6 weeks
  Objective surgical data such as operative time will be recorded between both groups and compared.
Objective surgical data such as estimated blood loss (EBL) | 6 weeks
  Objective surgical data such as estimated blood loss (EBL) will be recorded between both groups and compared.
Patient satisfaction (a decision scale and decision regret scale) | 3 months
  A decision regret scale will be administered to patients at 3 months postoperative, and scores will be compared between the two groups to assess if any difference in patient satisfaction exists.
Patient satisfaction (Patient Global Impression of Improvement (PGI-I) for Incontinence) | 3 months
  The PGI-I will be administered to all patients at 3 months to assess patient satisfaction with the procedure performed; any differences between groups in patient satisfaction will be assessed with this outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela E Halder, MD, MPH, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
Minimum necessay IPD will be shared with other researchers if trial is expanded to multiple sites.
Supporting Information: Study Protocol, SAP, Analytic Code